CLINICAL TRIAL: NCT01982812
Title: A Safety and Feasibility Study of Enteral Levetiracetam vs. Phenobarbital for Seizure Control in Pediatric Cerebral Malaria
Brief Title: A Safety and Feasibility Study of Enteral LVT vs. Standard of Care for Seizure Control in Pediatric CM
Acronym: LVT2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gretchen Birbeck, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7R01NS074409-02 (NIH); R01NS074409 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Seizure; Epilepsy; Cerebral Malaria
MeSH Terms: conditions — Seizures; Epilepsy; Malaria, Cerebral | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Levetiracetam (Experimental): Oral Levetiracetam administered by NG tube.
  Interventions: Drug: Oral Levetiracetam
- Standard AED (Active Comparator): Standard AED regimen
  Interventions: Drug: Standard AED

INTERVENTIONS:
Drug: Oral Levetiracetam — liquid, 40 mg/kg loading dose and 30mg/kg every 12 hours via nasogastric tube for 3 days
  Other Names: Keppra
  Arms: Oral Levetiracetam
Drug: Standard AED — Active comparitor, Standard AED
  Other Names: Standard regimen of AED therapy
  Arms: Standard AED

SUMMARY:
Pediatric cerebral malaria (CM) affects more than 3 million children each year killing ~20% and leaving one third of survivors with long term neurologic and psychiatric sequelae. Seizures occur commonly with CM and are associated with an increased risk of death and neuropsychiatric disabilities. In this Malawi-based, safety and feasibility study of enteral levetiracetam in pediatric CM, the investigators will lay the groundwork for future efficacy studies aimed at improving seizure control and ultimately decreasing the neurologic morbidity of pediatric CM.

DETAILED DESCRIPTION:
Cerebral malaria (CM) affects ~3 million children each year, primarily in sub-Saharan Africa. Antimalarial medications can rapidly clear P. falciparum parasites, but mortality rates remain high (12-25%). Survivors do not escape unscathed--~30% experience neurologic sequelae including epilepsy, behavioral disorders and gross neurologic deficits. Acute seizures occur commonly in CM and are associated with higher neurologic morbidity and mortality. Seizure management in malaria endemic regions is challenging because the available antiepileptic drugs (AED) induce respiratory suppression and assisted ventilation is unavailable. More optimal seizure control may improve neurologic outcomes in pediatric CM survivors, especially if the medication used is affordable and can be delivered safely and easily in resource limited settings. The investigators conducted a dose- escalation study detailed elsewhere (NCT01660672) to determine the optimal dose for use in this safety and feasibility study of enteral levetiracetam (LVT) for seizure control in children with CM and seizures admitted to Queen Elizabeth Central Hospital in Blantyre, Malawi. Enteral LVT given via nasogastric tube (NGT) rather than an intravenous (IV) formulation will be used since LVT has excellent enteral bioavailability and IV formations are not affordable in most malaria-endemic regions. LVT 40mg/kg followed by 30mg per kg Q12 hourly. Children admitted with cerebral malaria and seizures will be randomized to LVT vs. standard of care with phenobarbital as needed comparing seizure control, safety, and neurological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Comatose with Blantyre Comas Score ≤ 2
* P. falciparum parasitemia via thick blood film or rapid diagnostic test
* Active seizure in past 24 hours

Exclusion Criteria:

* Serum creatinine > 2mg/dL
* Pre-admission/concomitant treatment with antiretroviral medications for HIV (ARVs), antituberculous treatments(ATTs), or chronic use of any other enzyme-inducing medications

Ages: 24 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L Birbeck, M.D., Principal Investigator — University of Rochester
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
After the finding have been published, the de-identified study data will be available to other researchers on request pending a review of their plans for using the data.

REFERENCES:
- [Derived] Birbeck GL, Herman ST, Capparelli EV, Dzinjalamala FK, Abdel Baki SG, Mallewa M, Toto NM, Postels DG, Gardiner JC, Taylor TE, Seydel KB. A clinical trial of enteral Levetiracetam for acute seizures in pediatric cerebral malaria. BMC Pediatr. 2019 Nov 1;19(1):399. doi: 10.1186/s12887-019-1766-2. PMID 31672143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized consecutive, eligible consented children with cerebral malaria during two recruitment periods--January to June 2014 and 2015,
Groups:
- Comparison Group: 2014: Children randomized to routine care who then recieved 20mg/kg phenobarbital with additional doses at the managing clinicians discretion
  2015: Children randomized to routine care will phenobarbital given at the discretion of the managing clinician but with a max od 20mg/kg load
Period: Overall Study
Arm/Group | Oral Levetiracetam | Comparison Group
Started | 23 | 21
Completed | 22 | 11
Not Completed | 1 | 10
Not completed — Death | 1 | 5
Not completed — Adverse Event | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Levetiracetam | Standard AED | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 21 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 41.4 (10.6) | 41.8 (16.7) | 41.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 13 | 7 | 20
Race/Ethnicity, Customized [Number; unit: participants] — Everyone in this Malawian study population was a black African
  participants
    African | 23 | 21 | 44
cerebral malaria retinopathy (present) [Number; unit: participants]
  retinopathy positive | 16 | 12 | 28
  retinopathy negative | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Minutes With Seizure on EEG
Description: Comparing LVT to standard AED the number of minutes spent in seizure per cEEG in the 72 hours after treatment allocation.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: minutes with seizure
Arm/Group | Oral Levetiracetam | Comparison Group
Number analyzed (Participants) | 23 | 21
minutes with seizure | 165.2 (265.9) | 464.8 (639.3)

2. Secondary Outcome: Required Additional AED
Description: Additional AEDs required (including for breakthrough seizures in LVT group) during admission for seizure control (yes/no)
Time Frame: 7 days
Measure: Number; unit: Participants requiring additional AEDs
Arm/Group | Oral Levetiracetam | Comparison Group
Number analyzed (Participants) | 23 | 21
Participants requiring additional AEDs | 18 | 18

3. Secondary Outcome: Mean Time From Admission to BCS >/= 4
Description: The mean time in hours from admission until the subject reaches Blantyre Coma Scale of greater than or equal to 4. Participants who died are excluded from this analysis.
  The Blantyre Coma Score has ranges from 0-5 based upon the a sum of the following 3 domains- Eye movement
  1 - Watches or follows 0 - Fails to watch or follow
  Best motor response 2 - Localizes painful stimulus 1 - Withdraws limb from painful stimulus 0 - No response or inappropriate response
  Best verbal response 2 - Cries appropriately with pain, or, if verbal, speaks
  1 - Moan or abnormal cry with pain 0 - No vocal response to pain
Time Frame: 7 days
Population: Comparing mean time to coma resolution in hours among survivors
Measure: Mean (Standard Deviation); unit: hours of coma from admission
Arm/Group | Oral Levetiracetam | Comparison Group
Number analyzed (Participants) | 22 | 16
hours of coma from admission | 35.4 (29.0) | 34.6 (27.8)

4. Secondary Outcome: Sequelae
Description: Neurologic outcome in 3 categories--
  1. Neurologically intact at discharge
  2. Neurologic sequelae at discharge--specifically new sensory or motor deficits, ongoing seizures, or behavioral abnormalities based upon a physician examination at discharge
  3. Died during admission, never discharged
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Oral Levetiracetam | Comparison Group
Number analyzed (Participants) | 23 | 21
participants
  Neurologically intact at discharge | 19 | 14
  Neurologic sequelae at discharge | 3 | 2
  Died during admission | 1 | 5

ADVERSE EVENTS:
Time Frame: 1 month post enrollment
Arm/Group | Oral Levetiracetam | Comparison Group
Serious Adverse Events (participants affected / at risk) | 5/23 | 8/21
Other Adverse Events (participants affected / at risk) | 15/23 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Levetiracetam (N=23) | Comparison Group (N=21)
death (Nervous system disorders) | 1 (1) | 5 (5) — Died with respiratory then cardiac failure as is typical of death in pediatric cerebral malaria
elevated AST (Hepatobiliary disorders) | 3 (4) | 2 (2) — laboratory assessment at 24 hours, 7 days and 1 month post randomization
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — Persistent or worsening thrombocytopenia
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Based upon creatinine
respiratory suppression or aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Anemia (persistent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
elevated ALT (Hepatobiliary disorders) | 0 (0) | 0 (0) — laboratory assessment at 24 hours, 7 days and 1 month post randomization
elevated alkaline phosphatase (Hepatobiliary disorders) | 0 (0) | 0 (0) — laboratory assessment at 24 hours, 7 days and 1 month post randomization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Levetiracetam (N=23) | Comparison Group (N=21)
myoclonus (Nervous system disorders) | 1 (1) | 0 (0) — myoclonic jerks while fully awake
Anemia with persistent low retics (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — At 30 days post d/c
Increased AST (Hepatobiliary disorders) | 5 (7) | 7 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
elevated platelet count (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Decreased reticulocyte count (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Abnormal ECG (Cardiac disorders) | 0 (0) | 1 (1)
Excess sedation (Nervous system disorders) | 0 (0) | 1 (1)
Increased ALT (Hepatobiliary disorders) | 4 (4) | 4 (7)
Increased alkaline phosphotase (Hepatobiliary disorders) | 3 (3) | 5 (7)
Increased potassium (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Increased chloride (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
increased phosphate (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
increased calcium (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No